CLINICAL TRIAL: NCT00656968
Title: Sequential Versus Concomitant Therapy for Helicobacter Pylori Infection
Brief Title: Comparison of Sequential or Concomitant Therapy for Helicobacter Pylori Infection
Acronym: 960025
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU-IRB00003151; VGHKS95-CT3-11 (Other Grant/Funding Number: KaohsiungVGH)
Record Dates: First submitted 2008-01-03; First posted 2008-04-14 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Helicobacter Infection
Keywords: peptic ulcer disease; gastric cancer; therapeutics
MeSH Terms: conditions — Helicobacter Infections; Peptic Ulcer; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10-day concomitant therapy (Active Comparator): esomeprazole and amoxicillin and clarithromycin and metronidazole for 10 days
  Interventions: Drug: 10-day concomitant therapy
- 10-day sequential therapy (Experimental): esomeprazole and amoxicillin for 5 days, followed by esoprazole and clarithromycin and metronidazole for 5 more days
  Interventions: Drug: 10-day sequential treatment

INTERVENTIONS:
Drug: 10-day sequential treatment — esomeprazole (40 mg daily) from day 1 to day 10, amoxicillin (1 g, bid) from day 1 to day 5, clarithromycin (500 mg, bid) from day 6 to day 10, metronidazole (500 mg, bid) from day 6 to day 10
  Other Names: Nexium-based sequential therapy
  Arms: 10-day sequential therapy
Drug: 10-day concomitant therapy — esomeprazole (40 mg, bid) from day 1 to day 10, amoxicillin (1 g, bid) from day 1 to day 10, clarithromycin (500 mg, bid) from day 1 to day 10, metronidazole (500 mg, bid) from day 1 to day 10
  Other Names: Nexium-based quadruple therapy
  Arms: 10-day concomitant therapy

SUMMARY:
Helicobacter pylori is a bacteria that infects the lining of the stomach and is associated with ulcers. Helicobacter pylori may also increase the long-term risk of developing certain forms of gastric cancer. Curing this infection generally requires that patients take 2 or more antibiotic medications and a stomach acid suppressing medication for about two weeks. Current treatments do not always cure the infection and a new treatment is being tested in this study. The drugs involved in the new 4 drug treatment have been widely used for treatment of this infection. It remains unknown what is the best and most cost effective way to give them. This study will compare three different ways of using these drugs.

Subjects must have active Helicobacter pylori infection in order to participate in this study.

DETAILED DESCRIPTION:
The purpose of this study is to compare different methods of giving combination drug therapy for treating Helicobacter pylori infection of the stomach. The entire study will last less than 2 years. Each subject will be participating in the study for approximately 60 days.

A total of 360 subjects will be asked to participate in this study.

Before participating in this study, subject's must have undergone to confirm the presence and to assess the susceptibility of Helicobacter pylori. Qualified subjects will receive 4 drugs which are to be taken as part of the study treatment: an acid suppressing drug (name), amoxicillin, clarithromycin and metronidazole. The doses are 1 grams of amoxicillin, 40 mg of esomeprazole (Nexium), 500 mg of metronidazole and 250 mg of clarithromycin. Each drug will be given twice a day to be taken twice a day with the morning and evening meals. Subjects will receive one of three different combinations. The choice of which will be randomly chosen by the use of a computer program. The regimes are: all 4 drugs daily for 5 days, all 4 drugs daily for 10 days, and two drugs (esomeprazole and amoxicillin) for 5 days then all for drugs for 5 additional days.

Subjects will be asked to return within 4 days after completion of the treatment to evaluate how they did with the drugs. They will be asked bring back all unused medication and the bottles or containers that the medicine was packaged in. Your medication use and tolerance to the study drugs will be assessed. The treatment portion of the study will be complete at this point.

Evaluation of the effect of the treatment will take place 4-6 weeks after the end of therapy. Subjects will come back to the study site and will have a UBT or repeat endoscopy, if clinically indicated to verify that the Helicobacter pylori has been cured. Subjects will be asked not to take antibiotics or any other drugs that may affect the outcome of the breath test used to confirm that the treatment was successful.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 18 to 75 years inclusively.
* Mental and legal ability to give a written informed consent.
* Active H. pylori infection.

Exclusion Criteria:

* Previous surgery of the stomach such as partial gastrectomy.
* Use of antibiotics within the preceding 30 days.
* Regular use of bismuth compounds (>3 times per week) in the 30 days before enrollment.
* Presence of serious medical condition(s) precluding participation or endoscopy with biopsy.
* Use of concomitant medication(s) known to interact with study medication.
* Presence of Zollinger-Ellison Syndrome.
* Pregnancy or lactation.
* Allergy to any of the study medications.
* Contraindication(s) to the use of any of the study drugs.
* Participation in a clinical trial within the last 30 days.
* Unwillingness to abstain from alcoholic beverages.
* Patients taking other medications including warfarin, antipsychotics, or chronic NSAIDs will also be excluded. Aspirin at a dose not more than 325 mg/day will be permitted.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Kuan Liu, MD, PhD, Study Chair — Kaohsiung Medical Univestity; David Y Graham, MD, Study Chair — Baylor College of Medicine; Antone R Opekun, PA-C, Study Director — Baylor College of Medicine; Deng-Chyang Wu, MD PhD, Principal Investigator — Kaohsiung Medical University
Locations (2):
- Taiwan (2):
  - Chung-Ho Hospital, Kaohsiung, Taiwan
  - Kaohsiung Veterans General Hospital, Kaohsiung City

REFERENCES:
- [Background] Francavilla R, Lionetti E, Castellaneta SP, Magista AM, Boscarelli G, Piscitelli D, Amoruso A, Di Leo A, Miniello VL, Francavilla A, Cavallo L, Ierardi E. Improved efficacy of 10-Day sequential treatment for Helicobacter pylori eradication in children: a randomized trial. Gastroenterology. 2005 Nov;129(5):1414-9. doi: 10.1053/j.gastro.2005.09.007. PMID 16285942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We surveyed patients who visited the gastroenterological clinic of Kaohsiung Medical University Hospital (KMUH), Kaohsiung Veteran General Hospital (KVGH). A total of 232 H. pylori-infected patients were randomly assigned to sequential (n = 117) or concomitant (n = 115) therapies.
Groups:
- Concomitant Therapy (A): esoprazole (40 mg, bid), amoxicillin (1 g, bid), clarithromycin (500 mg, bid) and metronidazole (500 mg, bid) for 10 days
- Sequential Therapy (B): esoprazole (40 mg, bid) from day 1 to day 10, amoxicillin (1 g, bid) from day 1 to day 5, clarithromycin (500 mg, bid) from day 6 to day 10, and metronidazole (500 mg, bid) from day 6 to day 10
Period: Overall Study
Arm/Group | Concomitant Therapy (A) | Sequential Therapy (B)
Started | 115 | 117
Completed | 115 | 117
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Therapy (A) | Sequential Therapy (B) | Total
Number analyzed (Participants) | 115 | 117 | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 99 | 197
  >=65 years | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.3) | 51.7 (12) | 51.74 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 56 | 111
  Male | 60 | 61 | 121
Region of Enrollment [Number; unit: participants]
  Taiwan | 115 | 117 | 232

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: Evaluate eradication outcome by endoscopy urease test and histology or urea breath test
Time Frame: one month after finishing study drugs
Measure: Number; unit: participants
Arm/Group | Concomitant Therapy (A) | Sequential Therapy (B)
Number analyzed (Participants) | 115 | 117
participants | 92 | 95

2. Primary Outcome: Number of Participants Who Had Good Drug Compliance
Description: Good drug compliance is defined as taking equal to or more than 80% of eradication medicines
Time Frame: one month after finishing test therapy
Measure: Number; unit: participants
Arm/Group | Concomitant Therapy (A) | Sequential Therapy (B)
Number analyzed (Participants) | 115 | 117
participants | 106 | 104

ADVERSE EVENTS:
Arm/Group | Concomitant Therapy (A) | Sequential Therapy (B)
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/117
Other Adverse Events (participants affected / at risk) | 31/115 | 36/117
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Therapy (A) (N=115) | Sequential Therapy (B) (N=117)
bad taste (Gastrointestinal disorders) | 18 (18) | 12 (12) — Patients had taste perversion.
Dizziness (Nervous system disorders) | 13 (13) | 10 (10) — Patients had dizziness discomforts.
Fatigue (Nervous system disorders) | 5 (5) | 13 (13)
Headache (Nervous system disorders) | 5 (5) | 5 (5)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No